CLINICAL TRIAL: NCT03408483
Title: Quadratus Lumborum Block Versus Control for Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Promil Kukreja, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300000836
Record Dates: First submitted 2017-12-19; First posted 2018-01-24 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Total Hip Arthroplasty
Keywords: Quadratus Lumborum Block
MeSH Terms: interventions — NOP-bolus regimen; Bupivacaine; Epinephrine; Standard of Care; Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: In this randomized controlled study we aim to compare QLB (intervention) with control (no intervention) group in patients undergoing THA with regard to the VAS pain scores (at PACU arrival & dischage,12, 24 & 36 hours), duration of analgesia, time to first opioid medication, physical therapy evaluations, time to discharge, and surgeon and patient satisfaction scores.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- quadratus lumborum block (QLB) (Experimental): * Patients will be placed in the lateral decubitus position w/non-operative side recumbent. Pillow or blankets will be placed btw patient's lower extremities. Standard noninvasive monitors applied, and oxygen administered via nasal cannula. Parenteral midazolam and fentanyl titrated to patient comfort.
  * Standard skin sterilization, prepping and draping will be applied to the area. Under ultrasound guidance, needle will be advanced to anterior border of quadratus lumborum muscle. After negative aspiration, a bolus of 30 mL of 0.25% bupivacaine with 1:400,000 epinephrine will be injected in 5 mL aliquots.
  * After QLB is placed, patients will have THA under spinal anesthesia.
  Interventions: Drug: Quadratus Lumborum Block (QLB)
- Standard of Care (Active Comparator): * Patients will be placed in the lateral decubitus position with non-operative side recumbent. A pillow or blankets placed between patient's lower extremities. Standard noninvasive monitors applied, and oxygen administered via nasal cannula. Parenteral midazolam and fentanyl titrated to patient comfort.
  * Standard skin sterilization, prepping and draping applied to the area. Ultrasound probe used to identify quadratus lumborum muscle. No local anesthetic injected.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Quadratus Lumborum Block (QLB) — Under ultrasound guidance, the needle will be advanced to the posterior border of the quadratus lumborum muscle. After negative aspiration, a bolus of 40 mL of 0.25% bupivacaine with 1:400,000 epinephrine will be injected in 5 mL aliquots, ensuring proper placement of needle tip and appropriate spread of local anesthetic.
  Other Names: bolus; bupivacaine; epinephrine; aliquots
  Arms: quadratus lumborum block (QLB)
Drug: Standard of Care — This is currently the standard of care, no local anesthetic will be injected. Pain will be managed with parenteral and oral medication.
  Other Names: parenteral opioid; oral opioid
  Arms: Standard of Care

SUMMARY:
Peripheral nerve blocks for joint and extremity surgeries have long been proven to provide effective post-operative analgesia. Of these surgeries, total hip arthroplasty (THA) remains one of the most common orthopedic procedures in the United States with approximately 300,000 operations performed annually. At our institution, post-operative analgesia in these patients is primarily provided through parenteral and oral opioid medications. Quadratus lumborum blocks (QLB) have been described and implemented for various surgical procedures including caesarean and laparoscopic ovarian surgery. Recently, there has been increasing interest in the efficacy of quadratus lumborum blocks for THA. Currently, case reports have established a precedent regarding the efficacy of the QLB for THA in providing superior analgesia and decreasing visual analog pain scores (VAS), but randomized trials are still lacking. The goal of this study is to compare pain scores (VAS), opioid consumption, physical therapy scores, and patient and surgeon satisfaction in patients that receive QLB versus no peripheral nerve blockade in patients undergoing THA. The results of this study have the potential to change standard of care for patients undergoing THA.

DETAILED DESCRIPTION:
Currently, regional anesthesia techniques for total hip arthroplasty are limited. Fascia iliac blocks have been employed to provide analgesia for hip surgeries with blockade of the femoral, lateral femoral cutaneous, and obturator nerves via injection of local anesthetic in the iliacus fascia. In addition, lumbar plexus blocks have also been employed for post-operative analgesia, but the complexity of the block is high, and complications including epidural anesthesia are not infrequent. The quadratus lumborum block is an abdominal truncal block in which local anesthetic is deposited into the thoracolumbar fascia or the quadratus lumborum muscle itself with the goal of providing analgesia to the ipsilateral T6 - L1 sensory dermatomes. It has already been demonstrated to provide effective post-operative analgesia for certain abdominal and pelvic surgeries, but its use in total hip arthroplasty is limited to case reports.

The block is accomplished by identifying the quadratus lumborum muscle, which originates from iliac crest and iliolumbar ligament, and inserted on transverse processes of upper four lumbar vertebrae and posterior border of the 12th rib. Local anesthetic is then deposited at the anterior, posterior or middle thoracolumbar fascia, or intramuscularly, depending on the technique used. Cadaveric studies8 have demonstrated dye spread to the lumbar nerve roots and nerves within the transversus abdominis plane (TAP). Carney et al9 described a "posterior TAP" block, now known to be synonymous with QLB, that demonstrated contrast spread to the thoracic paravertebral space from T5-L1. Case reports have described analgesia in the corresponding sensory dermatomes after QLB4, and have demonstrated efficacy in patient undergoing THA. The QLB block has potential to cover lateral femoral cutaneous nerve, femoral nerve, obturator nerve and portions of lumbar plexus.

This study has been designed to investigate the efficacy of the quadratus lumborum block as a primary method of providing post-operative analgesia in patients undergoing THA. Previous trials have demonstrated the effectiveness of the block for abdominal and pelvic surgeries, and case reports have shown its applicability in hip arthroplasty. In this randomized controlled study we aim to compare QLB (intervention) with control (no intervention) group in patients undergoing THA with regard to the VAS pain scores (at PACU arrival & discharge12, 24 & 36 hours), duration of analgesia, time to first opioid medication, physical therapy evaluations, time to discharge, and surgeon and patient satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing total hip arthroplasty
2. Adults 18 years of age and older
3. Patients with an American Society of Anesthesiology (ASA) physical status classification of I, II or III

Exclusion Criteria:

1. Patients with ASA physical status classification other than I, II, or III
2. Patients with allergies/intolerances to local anesthetic
3. Patients with pre-existing neurologic or anatomic deficits in the lower extremity on the side of the surgical site
4. Patients with coexisting coagulopathy
5. Patients that are pharmacologically anticoagulated will be excluded if placement of peripheral nerve block would be contraindicated according to ASRA (American Society for Regional Anesthesia) guidelines or if spinal anesthesia would be contraindicated according to guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Promil Kukreja, MD, PhD, Principal Investigator — UAB Department of Anesthesiology, Critical Care Division
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Kukreja P, MacBeth L, Sturdivant A, Morgan CJ, Ghanem E, Kalagara H, Chan VWS. Anterior quadratus lumborum block analgesia for total hip arthroplasty: a randomized, controlled study. Reg Anesth Pain Med. 2019 Oct 25:rapm-2019-100804. doi: 10.1136/rapm-2019-100804. Online ahead of print. PMID 31653800

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadratus Lumborum Block (QLB): * Patients will be placed in the lateral decubitus position w/non-operative side recumbent. Pillow or blankets will be placed btw patient's lower extremities. Standard noninvasive monitors applied, and oxygen administered via nasal cannula. Parenteral midazolam and fentanyl titrated to patient comfort.
  * Standard skin sterilization, prepping and draping will be applied to the area. Under ultrasound guidance, needle will be advanced to anterior border of quadratus lumborum muscle. After negative aspiration, a bolus of 30 mL of 0.25% bupivacaine with 1:400,000 epinephrine will be injected in 5 mL aliquots.
    * After QLB is placed, patients will have THA under spinal anesthesia.
  Quadratus Lumborum Block (QLB): Under ultrasound guidance, the needle will be advanced to the posterior border of the quadratus lumborum muscle. After negative aspiration, a bolus of 40 mL of 0.25% bupivacaine with 1:400,000 epinephrine will be injected in 5 mL aliquots, ensuring proper placement of needle
- Standard of Care: * Patients will be placed in the lateral decubitus position with non-operative side recumbent. A pillow or blankets placed between patient's lower extremities. Standard noninvasive monitors applied, and oxygen administered via nasal cannula. Parenteral midazolam and fentanyl titrated to patient comfort.
  * Standard skin sterilization, prepping and draping applied to the area. Ultrasound probe used to identify quadratus lumborum muscle. No local anesthetic injected.
  Standard of Care: This is currently the standard of care, no local anesthetic will be injected. Pain will be managed with parenteral and oral medication.
Period: Overall Study
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Started | 42 | 38
Completed | 36 | 35
Not Completed | 6 | 3
Not completed — Physician Decision | 3 | 3
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Three patients in each group were excluded for failed spinal anesthesia. Three patients were excluded in the Quadratus Lumborum Block group for missing data due to early discharge.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.61 (2.74) | 58.00 (2.06) | 58.305 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Using Visual Analog Scale (VAS) Scores
Description: The Visual Analogue Scale (VAS) is a psychometric response scale which is used in surveys/questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older:
  Rating - Pain Level
  0 - No Pain
  1-3 - Mild Pain (nagging, annoying, interfering little with *ADLs)
  4-6 - Moderate Pain (interferes significantly with ADLs)
  7-10 - Severe Pain (disabling; unable to perform ADLs)
  *ADL=Activities of Daily Living
Time Frame: Assessed between immediately postoperatively to 12 hours postoperatively
Population: Three patients in each group were excluded for failed spinal anesthesia. Three patients were excluded in the QLB group for missing data due to early discharge.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 36 | 35
units on a scale | 2.34 (0.46) | 3.33 (0.56)

2. Primary Outcome: Pain Scores Using Visual Analog Scale (VAS) Scores
Description: as for outcome 1
Time Frame: Assessed between immediately postoperatively to 24 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 36 | 35
units on a scale | 2.31 (0.37) | 4.06 (0.42)

3. Primary Outcome: Pain Scores Using Visual Analog Scale (VAS) Scores
Description: as for outcome 1
Time Frame: Assessed between immediately postoperatively to 48 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
units on a scale | 3.33 (0.43) | 4.11 (0.64)

4. Primary Outcome: Opioid Consumption (Oral Morphine Equivalents)
Description: Total oral morphine equivalent consumption calculated
Time Frame: from 24 hours to 48 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg of morphine equivalents
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
mg of morphine equivalents | 24.26 (4.48) | 40.52 (6.31)

5. Primary Outcome: Opioid Consumption (Oral Morphine Equivalents)
Description: Total oral morphine equivalent consumption calculated
Time Frame: immediately postoperatively to 24 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg of morphine equivalents
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
mg of morphine equivalents | 30.05 (3.80) | 47.14 (4.72)

6. Primary Outcome: Opioid Consumption (Oral Morphine Equivalents)
Description: Total oral morphine equivalent consumption calculated
Time Frame: immediately postoperatively to 48 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg of morphine equivalents
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
mg of morphine equivalents | 54.63 (8.25) | 90.76 (10.65)

7. Primary Outcome: Pain Scores Using Visual Analog Scale (VAS) Scores
Description: as for outcome 1
Time Frame: Immediately postoperatively to 12 hours postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 36 | 35
score on a scale | 2.34 (0.46) | 3.33 (0.56)

8. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction Score:
  Determined by patient interview conducted at the 24 hour Time Frame.
  The interview follows a script requesting current pain level based on a scale of 1-10:
  1 = very not satisfied 10 = very satisfied
  Patient satisfaction is subjective.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
score on a scale | 9.14 (0.28) | 7.46 (0.41)

9. Secondary Outcome: Hours to Hospital Discharge
Description: From time of the surgical procedure to the time of hospital discharge (measured in hours) up to 3 hours.
Time Frame: Maximum 96 Hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hours
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
hours | 53.17 (4.99) | 55.97 (3.78)

10. Secondary Outcome: Distance Ambulated
Description: Physical therapist documentation of ambulation distance measured in feet
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: feet
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
feet | 127.75 (17.33) | 106.69 (23.37)

11. Secondary Outcome: Distance Ambulated
Description: Physical therapist documentation of ambulation distance measured in feet
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: feet
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
Number analyzed (Participants) | 35 | 36
feet | 114.51 (10.39) | 100.85 (10.60)

ADVERSE EVENTS:
Time Frame: From baseline through 18 months
Description: Three patients in each group were excluded for failed spinal anesthesia. Three patients were excluded in the QLB group for missing data due to early discharge.
Arm/Group | Quadratus Lumborum Block (QLB) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03408483/Prot_SAP_000.pdf